CLINICAL TRIAL: NCT00306410
Title: The Prevalence of Vitamin D Deficiency and Effects of Vitamin D Supplementation in HIV-1 Infected Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIDI trial
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Vitamin D Deficiency; HIV Infections
Keywords: Vitamin D deficiency; HIV/AIDS; HAART; T-Lymphocytes, Regulatory; insulin resistance; bone density
MeSH Terms: conditions — Vitamin D Deficiency; HIV Infections; Acquired Immunodeficiency Syndrome; Insulin Resistance | interventions — Cholecalciferol

INTERVENTIONS:
Drug: colecalciferol

SUMMARY:
The purpose of this study is to determine the effect of normalization of vitamin D levels on bone density, immune and adipocyte function in HIV1-seropositive patients.

DETAILED DESCRIPTION:
Vitamin D deficiency is common in, especially black, HIV-seropositive patients. Vitamin D deficiency can be caused by lack of sunlight and/or insufficient vitamin D intake via diet. The HIV infection itself and antiretroviral therapy (ART) may also cause vitamin D deficiency. ART interferes with cytochrome p450 activity and as such might affect vitamin D metabolism.

Vitamin D has several important physiological functions such as 1. regulation of calcium and phosphate homeostasis, 2. immunomodulatory properties and 3. effects on adipocyte differentiation. Low vitamin D levels lead to decreased bone mineralization, eventually resulting in rachitis(children) or osteomalacia (in adults). In addition vitamin D deficiency leads to secondary hyperparathyroidism, which leads to even more bone matrix demineralization. In HIV infected persons the overall prevalence of osteopenia and osteoporoses is 14-84% and 0-45% respectively. Vitamin D has been suggested to play a role in HIV-associated bone disorders. The vitamin D status also affects the host defence in HIV patients; a significantly lower CD4 cell count has been found in patients with 1,25(OH)vitamin D deficiency. Furthermore, the influence of vitamin D on adipocyte differentiation and the effect of HAART on vitamin D levels might be relevant for changes in fat distribution and the development of insulin resistance as is seen days after initiation of HAART.

Vitamin D is metabolized in the body trough cytochrome P450 enzymes. HAART might interact with vitamin D metabolism on basis of CYP3A4, which plays an important role in clearance of most antiretroviral agents and also showed to be a vitamin D 24 and 25-hydroxylase in vitro. We hypothesize that PI's lead to lower 1a,25(OH)2D3 by suppressing 1a- and 25-hydroxylase activity.

The results of our pilot showed that 25(OH)D deficiency is common among HIV patients. Seen the diversity of functions of vitamin D, we hypothesize that it's beneficial for the patients to have a normal vitamin D status. Therefore, supplementation of vitamin D is warranted.

In this study we want to investigate if, despite the complex interaction between HAART/ HIV and vitamin D metabolism, supplementation of colecalciferol (2000 IU daily) will lead to normalization of the vitamin D levels. Furthermore, we want to study the effects of normalization of vitamin D levels on bone mineral density, immune and adipocyte function. Therefore we will do a prospective, randomized, double-blind, placebo-controlled vitamin D intervention study in vitamin D deficient HIV1-seropositive patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 jr
* able to give informed consent
* HIV seropositive diagnosed with standard techniques
* Hypovitaminoses D

Exclusion Criteria:

* Hypercalcemia: calcium levels >2.60 mmol/L
* Renal disorders: serum creatinine >2 times Upper limit of normal (ULN) (110 mmol/l)
* Liver disorders; elevation of ASAT or ALAT >5 x ULN. The ULNs are 40 IU/L and 45 IU/L for ASAT and ALAT, respectively.
* Pregnancy
* Drug or alcohol abuse
* Non compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2006-01; Study Completion 2007-07

PRIMARY OUTCOMES:
normalization of vitamin D levels at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: André JAM van der Ven, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] Madeddu G, Spanu A, Solinas P, Calia GM, Lovigu C, Chessa F, Mannazzu M, Falchi A, Mura MS, Madeddu G. Bone mass loss and vitamin D metabolism impairment in HIV patients receiving highly active antiretroviral therapy. Q J Nucl Med Mol Imaging. 2004 Mar;48(1):39-48. PMID 15195003
- [Background] Haug CJ, Aukrust P, Haug E, Morkrid L, Muller F, Froland SS. Severe deficiency of 1,25-dihydroxyvitamin D3 in human immunodeficiency virus infection: association with immunological hyperactivity and only minor changes in calcium homeostasis. J Clin Endocrinol Metab. 1998 Nov;83(11):3832-8. doi: 10.1210/jcem.83.11.5270. PMID 9814454
- [Background] Cozzolino M, Vidal M, Arcidiacono MV, Tebas P, Yarasheski KE, Dusso AS. HIV-protease inhibitors impair vitamin D bioactivation to 1,25-dihydroxyvitamin D. AIDS. 2003 Mar 7;17(4):513-20. doi: 10.1097/00002030-200303070-00006. PMID 12598771
- [Background] Mondy K, Powderly WG, Claxton SA, Yarasheski KH, Royal M, Stoneman JS, Hoffmann ME, Tebas P. Alendronate, vitamin D, and calcium for the treatment of osteopenia/osteoporosis associated with HIV infection. J Acquir Immune Defic Syndr. 2005 Apr 1;38(4):426-31. doi: 10.1097/01.qai.0000145352.04440.1e. PMID 15764959
- [Background] Holick MF. Vitamin D: important for prevention of osteoporosis, cardiovascular heart disease, type 1 diabetes, autoimmune diseases, and some cancers. South Med J. 2005 Oct;98(10):1024-7. doi: 10.1097/01.SMJ.0000140865.32054.DB. PMID 16295817